CLINICAL TRIAL: NCT07398560
Title: Adebrelimab Combined With Oral Etoposide for Elderly Patients and Patients With Poor Performance Status in Small Cell Lung Cancer: An Exploratory Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Third Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Liu Fang, Director, The Third Affiliated Hospital of Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-HLJ-015
Record Dates: First submitted 2026-01-25; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer; Oral etoposide; Elderly patients
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab Combined with Oral Etoposide (Experimental): Adebrelimab: 1200 mg, administered by intravenous infusion, once every 3 weeks, repeated until disease progression, unacceptable toxicity, or the patient has received a cumulative total of 2 years of adebrelimab treatment.
  Oral etoposide soft capsules: 75 mg, days 1-14, orally once daily, administered for 2 weeks followed by 1 week off.
  Investigators may administer prophylactic cranial irradiation at their discretion.
  Interventions: Drug: Adebrelimab; Drug: Oral etoposide soft capsules

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab: 1200 mg, administered by intravenous infusion, once every 3 weeks, repeated until disease progression, unacceptable toxicity, or the patient has received a cumulative total of 2 years of adebrelimab treatment.
Drug: Oral etoposide soft capsules — Oral etoposide soft capsules: 75 mg, days 1-14, orally once daily, administered for 2 weeks followed by 1 week off.

SUMMARY:
This is a multicenter, single-arm, exploratory clinical study designed to observe and evaluate the efficacy and safety of adebrelimab combined with oral etoposide for elderly patients and patients with poor performance status in small cell lung cancer.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, exploratory clinical study planned to enroll 47 patients, aiming to evaluate the efficacy and safety of adebrelimab combined with oral etoposide for elderly patients and patients with poor performance status in small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Extensive-stage or locally advanced small cell lung cancer at initial diagnosis.
2. Confirmed by pathological histology/cytology combined with imaging.
3. ECOG PS 2-3 or age ≥65 years.
4. If a large number of comorbidities exist: ① mild failure or cachexia; ② mild bone marrow reserve dysfunction; ③ mild cardiovascular, liver, or kidney dysfunction, or dysfunction of other important organs; ④ mild infection, provided anti-infection treatment is administered; ⑤ mild water-electrolyte or acid-base imbalance, provided symptomatic treatment is given; ⑥ incomplete gastrointestinal obstruction caused by tumors; ⑦ other mild contraindications to anti-tumor therapy, if the investigator determines that the patient can be enrolled (reference: Modern Oncology, 3rd Edition, Tang Zhaoyou, Antitumor Drug Therapy, Contraindications), then patients with ECOG PS 0-1 and age <65 are allowed.
5. Has measurable tumor target lesions (meeting RECIST 1.1 criteria).
6. Expected survival > 3 months.
7. The functions of major organs meet the following requirements (excluding the use of any blood components and cell growth factors during the screening period):

   1. Complete blood count (without blood transfusion or use of hematopoietic growth factors to correct the condition within 14 days): Hemoglobin (Hb) ≥90 g/L; Absolute neutrophil count (ANC) ≥1.5×10^9 /L; Platelets (PLT) ≥100×10^9 /L; White blood cell count (WBC) ≥3.0×10^9 /L.
   2. Biochemical tests: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (for patients with liver metastases, ≤ 5×ULN); serum total bilirubin (TBIL) ≤ 1.5×ULN (for subjects with Gilbert's syndrome, ≤ 3×ULN); serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance ≥ 50 ml/min.
   3. Coagulation function: Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤1.5×ULN.
   4. Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.
8. Women of childbearing age must have a negative pregnancy test (βHCG) before starting treatment. Women of childbearing age and men (who have sexual relations with women of childbearing age) must agree to use effective contraception continuously during the treatment and for 6 months after the last dose.
9. The patient voluntarily joined this study and signed the informed consent form.

Exclusion Criteria:

1. Within the past 2 years, having had or currently having other malignant tumors, except for cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, superficial or non-invasive bladder cancer, etc.
2. Active tuberculosis infection.
3. Individuals with uncontrolled or symptomatic brain metastases, a history of poorly controlled psychiatric disorders, or severe intellectual or cognitive impairments.
4. Participants with active, known, or suspected autoimmune diseases, those with hypothyroidism requiring only hormonal replacement therapy, or those with skin conditions not requiring systemic treatment (such as vitiligo, psoriasis, or hair loss) can be included.
5. Pleural effusion, pericardial effusion, or ascites that cannot be controlled and require repeated drainage (patients whose effusion has been stable for 2 weeks or more after treatment can be enrolled).
6. Subjects with any of the following severe and/or uncontrolled diseases, including:

   1. Subjects with poorly controlled blood pressure (systolic >160 mmHg or diastolic >100 mmHg).
   2. Patients with ≥Grade 2 myocardial ischemia or myocardial infarction, severe arrhythmias (including QTc ≥450 ms in men, QTc ≥470 ms in women), and ≥Grade 2 congestive heart failure (New York Heart Association [NYHA] classification).
7. History of psychiatric medication abuse, alcoholism, or drug use.
8. Active hepatitis (for hepatitis B reference: HBsAg positive and HBV DNA test value greater than 500 IU/ml; for hepatitis C reference: HCV antibody positive and HCV viral load test value exceeding the upper limit of normal) human immunodeficiency virus (HIV, HIV 1/2 antibody) positive.
9. Severe bone marrow suppression is present.
10. Pregnant women or women who may be pregnant.
11. Patients who cannot comply with the trial protocol or cannot cooperate with follow-up.
12. Unable to swallow pills, malabsorption syndrome, or any condition that affects gastrointestinal absorption.
13. Researchers believe those who should not participate in this trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | up to 24 months
  Defined as the time from randomization to the first occurrence of disease progression with use of RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | up to 24 months
  Determined using RECIST v1.1 criteria, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.
Disease control rate | up to 24 months
  Disease Control Rate (DCR) is defined as the proportion of evaluable patients who achieve either an objective response (Complete or Partial Response) or maintain Stable Disease following a therapeutic intervention.
Overall Survival | up to 24 months
  Defined as the time from randomization to death from any cause.
Safety: Incidence of adverse events | up to 24 months
  Incidence of adverse events
Patient-Reported Outcomes (PROs) | Up to 24 months
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (Version 3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Liu, MD, Principal Investigator — The Third Affiliated Hospital of Harbin Medical University
Locations (1):
- The Third Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No